CLINICAL TRIAL: NCT02507297
Title: Sleep-Disordered Breathing and PAP in Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Leslie Swanson, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K23HL122461-01A1 (NIH)
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Sleep-disordered Breathing; Major Depressive Disorder
MeSH Terms: conditions — Sleep Apnea Syndromes; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PAP Group (Experimental): Positive airway pressure (PAP) delivered through an auto-titrating machine, to be used nightly
  Interventions: Device: Positive Airway Pressure (PAP)
- TAU Group (No Intervention): Treatment as usual through obstetrics

INTERVENTIONS:
Device: Positive Airway Pressure (PAP) — Positive airway pressure therapy entails use of a machine that blows pressurized room air through the airway (via a mask or nasal pillows, worn on the face) at a sufficient pressure to keep the upper airway open. The pressurized air acts as a splint. Participants randomized to PAP treatment will be offered PAP therapy using an auto-titrating device.
  Other Names: CPAP
  Arms: PAP Group

SUMMARY:
The goal of this study is to understand the contribution of sleep-disordered breathing (SDB) to one of the most common and debilitating adverse pregnancy outcomes, perinatal depression. The study is a randomized trial to test the efficacy of positive airway pressure (PAP) on sleep and depression symptoms in perinatal women. Participants will be pregnant women with depression and sleep-disordered breathing. Participants will be randomly assigned to receive either PAP therapy (PAP group) or treatment as usual within obstetrics (TAU group). Mood and sleep assessments will be completed at baseline, after 1 week of enrollment, and monthly thereafter through 12 weeks postpartum. Cortisol will be measured using saliva collection at baseline and again 8 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* 20-32 weeks gestation with a single, live fetus
* meet criteria for major depressive disorder per the Structured Clinical Interview for DSM-V (SCID)
* respiratory distress index (RDI; includes apneas, hypopneas, and respiratory effort-related arousals)≥5 per ambulatory assessment plus apnea symptoms (snoring, witnessed apnea, daytime sleepiness, sleep disturbance, snort arousals)
* stable dose (for ≥8 weeks) of a selective serotonin reuptake inhibitor (SSRI) OR free of all antidepressant medications past 4 weeks
* obstetrics care is at the University of Michigan, and the woman plans on delivering her baby at the University of Michigan

Exclusion Criteria:

* Diagnosis of bipolar disorder, posttraumatic stress disorder, schizophrenia or psychosis, dissociative disorders, eating disorder, obsessive-compulsive disorder, somatic symptom and related disorders, substance use disorder, panic disorder, agoraphobia per DSM-V
* diagnosis of, or suspicion for, narcolepsy or REM behavior disorder
* current SDB treatment; medical conditions for which PAP is contraindicated (e.g., pneumothorax, pneumocephalus, recent trauma, recent surgery)
* evidence of risk for drowsy driving (excessive daytime sleepiness plus history of motor vehicle accident or near miss due to sleepiness, fatigue, or inattention in past 12 months).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Swanson, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PAP Group | TAU Group
Started | 16 | 13
Completed | 15 | 12
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PAP Group | TAU Group | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.44 (5.39) | 27.31 (6.32) | 29.18 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 11 | 7 | 18
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Hamilton Rating Scale for Depression (HRSD) Score, Excluding the Sleep Items [Mean (Standard Deviation); unit: units on a scale] — Clinician-rated depression severity and symptoms, excluding the items which measure sleep. Total score range: 0-46. Higher scores represent more severe depression.
  units on a scale | 15.06 (3.87) | 14.69 (3.68) | 14.9 (3.73)
Edinburgh Postnatal Depression Scale (EPDS) Score, Minus the Sleep Item [Mean (Standard Deviation); unit: units on a scale] — Self-reported measure of depression symptoms and severity, minus the sleep item. Total scores range from 0 to 27; higher scores indicate more severe depression.
  units on a scale | 11.88 (3.79) | 14.15 (3.76) | 12.9 (3.89)
Pittsburgh Sleep Quality Index (PSQI) Score [Mean (Standard Deviation); unit: units on a scale] — Measure of sleep quality. Total scores range from 0 to 21. Higher scores indicate worse sleep quality.
  units on a scale | 9.63 (2.99) | 10.92 (3.12) | 10.21 (3.06)
Epworth Sleepiness Scale (ESS) Score [Mean (Standard Deviation); unit: units on a scale] — Measure of excessive daytime sleepiness. Scores range from 0 to 25. Higher scores indicate more daytime sleepiness.
  units on a scale | 12.44 (4.03) | 8.54 (4.16) | 10.69 (4.47)
Salivary cortisol [Mean (Standard Deviation); unit: nmol/L] — Salivary cortisol is a hormone produced by the adrenal gland. Values are in nmol/L; detectable assay range is 0.33 - 82.77 nmol/L. Higher values indicate higher levels of cortisol.
  nmol/L | 33.07 (6.89) | 33.02 (10.82) | 33.05 (8.69)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Rating Scale for Depression (HRSD) Score, Minus the Sleep Item
Description: Change in clinician-rated depression severity and symptoms, excluding the items which measure sleep. Total score range: 0-46. Higher scores represent more severe depression.
Time Frame: Baseline to 8 weeks after baseline, and at 12 weeks postpartum
Population: Data are not available for 3 participants of the 16 participants started in the PAP group at baseline to 8 weeks. Data are not available for 3 participants of the 16 participants started in the PAP group at baseline to 12 weeks and 2 participants of the 13 participants started in the TAU group at baseline to 12 weeks postpartum.
Measure: Mean (Standard Deviation); unit: change in score
Arm/Group | PAP Group | TAU Group
Number analyzed (Participants) | 13 | 13
change in score
  Baseline to 8 weeks after baseline | -7.62 (5.65) | -5.92 (3.47)
  Baseline to 12 weeks postpartum: number analyzed (Participants) | 13 | 11
  Baseline to 12 weeks postpartum | -8.21 (7.39) | -6.18 (6.51)
Statistical Analysis 1: Comparison: PAP Group vs TAU Group; Baseline to 8 weeks after baseline; Test type: Superiority; p = .367, t-test, 2 sided
Statistical Analysis 2: Comparison: PAP Group vs TAU Group; Baseline to 12 weeks postpartum; Test type: Superiority; p = .48, t-test, 2 sided

2. Secondary Outcome: Change in Edinburgh Postnatal Depression Scale Score
Description: Change in a self-report measure of depression symptoms and severity. Total scores range from 0 to 27; higher scores indicate more severe depression.
Time Frame: Baseline to 8 weeks after baseline, and at 12 weeks postpartum
Population: Data for the baseline to 12 weeks postpartum analysis are not available for 3 participants of the 13 participants started in the TAU group and for 2 participants of the 16 participants started in the PAP group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAP Group | TAU Group
Number analyzed (Participants) | 16 | 13
score on a scale
  Baseline to 8 weeks after baseline | -4.13 (3.11) | -2.23 (3.51)
  Baseline to 12 weeks postpartum: number analyzed (Participants) | 14 | 10
  Baseline to 12 weeks postpartum | -3.00 (3.88) | -5.00 (5.85)
Statistical Analysis 1: Comparison: PAP Group vs TAU Group; Baseline to 8 weeks after baseline; Test type: Superiority; p = .136, t-test, 2 sided
Statistical Analysis 2: Comparison: PAP Group vs TAU Group; Baseline to 12 weeks postpartum; Test type: Superiority; p = .324, t-test, 2 sided

3. Secondary Outcome: Change in Pittsburgh Sleep Quality Index Score
Description: Change in a measure of sleep quality. Total scores range from 0 to 21. Higher scores indicate worse sleep quality.
Time Frame: Baseline to 8 weeks after baseline, and at 12 weeks postpartum
Population: Data for 2 participants of the 16 participants started in the PAP group are not available in the baseline to 8 weeks after baseline analysis and data for 3 participants from the 13 participants started in the TAU group are not available in the baseline to 8 weeks after baseline analysis. Data from 3 participants from the 13 participants started in the TAU group and 2 participants of the 16 participants started in the PAP group are not available in the baseline to 12 weeks analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAP Group | TAU Group
Number analyzed (Participants) | 14 | 13
score on a scale
  Baseline to 8 weeks after baseline: number analyzed (Participants) | 14 | 10
  Baseline to 8 weeks after baseline | -1.64 (3.10) | -1.80 (4.16)
  Baseline to 12 weeks postpartum: number analyzed (Participants) | 14 | 10
  Baseline to 12 weeks postpartum | -1.29 (3.67) | -1.8 (4.16)
Statistical Analysis 1: Comparison: PAP Group vs TAU Group; Baseline to 8 weeks after baseline; Test type: Superiority; p = .916, t-test, 2 sided
Statistical Analysis 2: Comparison: PAP Group vs TAU Group; Baseline to 12 weeks postpartum; Test type: Superiority; p = .752, t-test, 2 sided

4. Secondary Outcome: Change in Epworth Sleepiness Scale (ESS) Score
Description: Change in a measure of excessive daytime sleepiness. Scores range from 0 to 25. Higher scores indicate more daytime sleepiness.
Time Frame: Baseline to 8 weeks after baseline, and at 12 weeks postpartum
Population: Data are not available for 2 participants of the 16 participants started in the PAP group at baseline to 8 weeks and 3 participants of the 13 participants started in the TAU group at baseline to 8 weeks. Data are not available for 2 participants of the 16 participants started in the PAP group at baseline to 12 weeks and 3 participants of the 13 participants started in the TAU group at baseline to 12 weeks postpartum.
Measure: Mean (Standard Deviation); unit: change in score
Arm/Group | PAP Group | TAU Group
Number analyzed (Participants) | 14 | 10
change in score
  Baseline to 8 weeks after baseline | -2.14 (4.14) | -1.00 (5.54)
  Baseline to 12 weeks postpartum | -2.14 (4.15) | -1 (5.54)
Statistical Analysis 1: Comparison: PAP Group vs TAU Group; Baseline to 8 weeks after baseline; Test type: Superiority; p = .568, t-test, 2 sided
Statistical Analysis 2: Comparison: PAP Group vs TAU Group; Baseline to 12 weeks postpartum; Test type: Superiority; p = .568, t-test, 2 sided

5. Secondary Outcome: Change in Salivary Cortisol
Description: Salivary cortisol is a hormone produced by the adrenal gland. Values are in nmol/L; detectable assay range is 0.33 - 82.77 nmol/L. Higher values indicate higher levels of cortisol.
Time Frame: Baseline to 8 weeks after baseline
Population: Data are not available for 4 participants of the 16 participants started in the PAP group and 3 participants of the 13 participants started in the TAU group.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | PAP Group | TAU Group
Number analyzed (Participants) | 12 | 10
nmol/L | -1.23 (7.23) | 1.38 (9.98)
Statistical Analysis 1: Comparison: PAP Group vs TAU Group; Test type: Superiority; p = .486, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization until participants reached 12 weeks postpartum (the final time point in the study).
Description: Participants were queried about adverse events each time they completed the clinical assessment (Hamilton Rating Scale for Depression). Adverse event information was also obtained from participants' medical records.
  Note that participants in the TAU group were not at risk for the adverse events related to positive airway pressure (PAP) treatment as they were not assigned to receive PAP treatment; these adverse events are denoted by a 0 in the denominator for at risk designation for TAU group.
Arm/Group | PAP Group | TAU Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 3/16 | 0/13
Other Adverse Events (participants affected / at risk) | 10/16 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP Group (N=16) | TAU Group (N=13)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0) — Hyperbilirubinemia in participant's infant requiring hospitalization of infant
Postpartum hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PAP Group (N=16) | TAU Group (N=13)
Skin irritation (Skin and subcutaneous tissue disorders) | 5 (5) | 0/0 (0) — Skin irritation specifically related to CPAP mask
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0/0 (0) — Dry mouth specifically related to CPAP usage
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/0 (0) — Nasal congestion specifically related to CPAP usage
Claustrophobia (Psychiatric disorders) | 2 (2) | 0/0 (0) — Claustrophobia when using CPAP mask
Insomnia (Nervous system disorders) | 2 (2) | 0/0 (0) — Insomnia specifically related to using CPAP or to in-lab sleep night (only PAP participants completed the in-lab sleep night)
Depression (Psychiatric disorders) | 4 (4) | 3 (3) — Worsening of depression from baseline
Diabetes mellitus (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) — Gestational diabetes
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Small for gestational age (infant) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Participant's infant was small for gestational age
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — Distress/anxiety in completing study questionnaires

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT02507297/Prot_SAP_000.pdf